CLINICAL TRIAL: NCT00422942
Title: An Open-label, Exploratory Study of the Pharmacokinetic and Pharmacodynamic Activity of MabThera in Combination With Methotrexate in Synovial Tissue and in Peripheral Blood of Patients With Active Rheumatoid Arthritis.
Brief Title: A Pharmacokinetic and Pharmacodynamic Study of MabThera (Rituximab) Plus Methotrexate in Patients With Rheumatoid Arthritis (RA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated after enrollment of 3 participants due to recruitment difficulties.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA19078
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: Methotrexate

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15
Drug: Methotrexate — 10-25mg po weekly

SUMMARY:
This single arm study will investigate the pattern of B cell depletion in synovial tissue and peripheral blood of patients with active RA, after MabThera (1000mg iv x 2 on days 1 and 15) + methotrexate (10-25mg/week po) treatment. The clinical efficacy and pharmacokinetic profile of MabThera after treatment and retreatment will also be investigated. The anticipated time on study treatment is 2+ years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients 18-80 years of age;
* RA for >=3 months;
* receiving outpatient treatment;
* failed treatment with >=1 DMARD (but not anti TNF or other biologic therapy);
* inadequate response to methotrexate, having taken and tolerated it for >=12 weeks, with a stable dose for >=4 weeks.

Exclusion Criteria:

* rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA;
* history of, or current, inflammatory joint disease other than RA, or other systemic autoimmune disorder;
* diagnosis of RA before the age of 16;
* bone/joint surgery within 12 weeks of study;
* prior use of anti-TNF or other biologic therapy, an anti-alpha 4 integrin, or any cell-depleting therapies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Methotrexate (MTX): Participants received rituximab 1000 milligrams (mg) via intravenous (IV) infusion on Days 1 and 15 and also on Days 169 and 183 (for those meeting retreatment criteria) or as needed (PRN) if retreatment criteria were not met; premedication with methylprednisolone (MP) 100 mg IV was administered at least 30 minutes prior to each rituximab infusion. Participants also received MTX 10-25 mg per week (mg/week; oral or parenteral) for up to 48 weeks and folate (greater than or equal to [≥]5 mg/week) given as either a single weekly dose or as divided dose for up to 48 weeks.
Period: Overall Study
Arm/Group | Rituximab + Methotrexate (MTX)
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study terminated by Sponsor | 3

BASELINE CHARACTERISTICS:
Groups:
- Rituximab + MTX: Participants received rituximab 1000 mg via IV infusion on Days 1 and 15 and also on Days 169 and 183 (for those meeting retreatment criteria) or PRN if retreatment criteria were not met; premedication with MP 100 mg IV was administered at least 30 minutes prior to each rituximab infusion. Participants also received MTX 10-25 mg/week (oral or parenteral) for up to 48 weeks and folate (≥5 mg/week) given as either a single weekly dose or as divided dose for up to 48 weeks.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Absolute B Cell Cluster Differential 19 Positive (CD19+) Counts in Synovial Tissues
Description: The change from baseline in absolute B cell (CD19+) counts at each visit calculated as (B cell count at visit minus B cell count at baseline) for synovial tissues.
Time Frame: Weeks 12, 24, and 36
Population: No participant data were analyzed. Study was terminated after enrollment of 3 participants as it was decided that it would not be appropriate to expose further participants to study drug since the objectives and data sought from this study had been published from other, independent sources and given the recruitment difficulties encountered.
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Absolute Counts of Cells Expressing CD20+ and CD22+ in Absolute B Cell (CD19+) Counts in Synovial Tissues
Description: The change in absolute counts of cells expressing the key B cell markers (CD20+ and CD22+) in absolute B cell (CD19+) counts in synovial tissues at Weeks 12, 24, and 36, relative to baseline.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in Absolute Counts of Cells Expressing CD20+ and CD22+ in Absolute B Cell (CD19+) Counts in Peripheral Blood
Description: The change in absolute counts of cells expressing the key B cell markers (CD20+ and CD22+) in absolute B cell (CD19+) counts in peripheral blood at Weeks 4,12, 24, 36, and 48, relative to baseline.
Time Frame: Weeks 4,12, 24, 36, and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Levels of Key Cytokines (Interleukin [IL]-1beta [β], Tumor Necrosis Factor [TNF]-Alpha [α], IL-4, IL-6, IL-10, and IL-13) in Blood (Serum)
Description: The change in levels of key cytokines (IL-1β, TNF-α, IL-4, IL-6, IL-10, and IL-13) in blood (serum) on Days 15 and 183 and at Weeks 4, 12, 24, 36, and 48, relative to baseline.
Time Frame: Days 15 and 183 and Weeks 4, 12, 24, 36, and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Levels of Key Cytokines in (IL-1β, TNF-α, IL-6, and IL-10) in Synovial Tissues
Description: The change in levels of key cytokines in (IL-1β, TNF-α, IL-6, and IL-10) in synovial tissues at Weeks 12, 24, and 36, relative to baseline.
Time Frame: Weeks 12, 24, and 36
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Myelocytomatosis Oncogene (C-myc) and BCL2-associated X Protein (BAX) in Peripheral Blood
Description: The change in ribonucleic acid (RNA) expression of markers of apoptosis (C-myc and BAX) in peripheral blood at Days 15 and 183, relative to baseline.
Time Frame: Days 15 and 183
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

7. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Percent (20%) 50%, and 70% (ACR20/50/70) Response
Description: ACR20/50/70 response is greater than or equal to (≥) 20%, 50%, or 70% improvement, respectively, in tender joint count (TJC) and swollen joint count (SJC); and improvement in at least 3 of 5 remaining ACR core measures: patient assessment of pain; patient global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Week 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joint Count (DAS28) Erythrocyte Sedimentation Rate (ESR) Score
Description: The change in DAS28-ESR at Weeks 12, 24, 36, and 48, relative to baseline. DAS28-ESR was calculated from SJC and TJC using 28-joint count, ESR (millimeters per hour [mm/hour]) and patient global assessment of disease activity (participant-rated arthritis activity assessment). Total score range: 0-9.4, higher score equals (=) more disease activity. DAS28-ESR less than or equal to (≤) 3.2 implied low disease activity and greater than (>)3.2 to 5.1 implied moderate to high disease activity, and DAS28-ESR <2.6 = remission.
Time Frame: Weeks 12, 24, 36, and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants Achieving Response by European League Against Rheumatism (EULAR) Category
Description: The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 ≤ 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤ 5.1 or change from baseline >0.6 to ≤ 1.2 with DAS28 ≤ 5.1; non-responders: change from baseline ≤ 0.6 or change from baseline >0.6 and ≤ 1.2 with DAS28 >5.1.
Time Frame: Weeks 24, 36, and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in ACR Core Set
Description: The changes from baseline in the ACR core set parameters at Week 48. Change from baseline to Week 48 over time in ACR core set: SJC, TJC, physician's global assessment of disease activity, patient's global assessment of disease activity, patient's assessment of pain, HAQ, ESR, and CRP. ACR20/50/70 response: ≥20%/50%/70% improvement in SJC; ≥20%/50%/70% improvement in TJC; and ≥20%/50%/70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; physician's global assessment of disease activity, participant's assessment of disease activity, participant assessment of functional disability via a HAQ, and CRP at each visit.
Time Frame: Week 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS)
Description: mTSS = sum of erosion and Joint Space Narrowing (JSN) scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change: scores at observation minus score at baseline. An increase in mTSS from baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline in Erosion Score
Description: Changes from baseline in modified Sharp radiographic erosion score from baseline to Weeks 24 and 48. The change in score at week X (where X=Week 24 or Week 48, as appropriate) calculated as: Change = week X score minus screening score.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in Joint Space Narrowing (JSN) Score
Description: Changes from baseline in modified Sharp radiographic JSN score from baseline to Weeks 24 and 48. The change in score at week X (where X=Week 24 or Week 48, as appropriate) calculated as: Change = week X score minus screening score.
Time Frame: Weeks 24 and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

14. Primary Outcome: Change From Baseline in Absolute B Cell CD19+ Counts in Peripheral Blood
Description: The change from baseline in absolute B cell (CD19+) count at each visit calculated as (B cell count at visit minus B cell count at baseline) for peripheral blood.
Time Frame: Weeks 4, 12, 24, 36, and 48
Population: as for outcome 1
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Rituximab + MTX
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Study terminated after enrollment of 3 participants due to recruitment difficulties and since the objectives and data under study had been published from other, independent sources it was not appropriate to expose further participants to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.